CLINICAL TRIAL: NCT04202952
Title: A Phase Ib/IIa, Single Center, Randomized, Open, Sofosbuvir-controlled, Multiple Ascending Dose Study to Access the Tolerability， Pharmacokinetics and Pharmacodynamics of HEC110114 Tablets in HCV-infected Subjects
Brief Title: The Tolerability, Pharmacokinetics and Pharmacodynamics Study of HEC110114 Tablets in HCV-infected Subjects
Acronym: HEC110114
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEC110114-P-02
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2019-12

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 600 mg multiple doses (Experimental): Subjects receiving 600 mg HEC110114 tablet (N=6) or sofosbuvir tablets(N=2) once daily (q.d.) for 3 days
  Interventions: Drug: HEC110114 Tablet; Drug: Sofosbuvir Tablet
- 800 mg multiple doses (Experimental): Subjects receiving 800 mg HEC110114 tablet (N=6) or sofosbuvir tablets(N=2) once daily (q.d.) for 3 days
  Interventions: Drug: HEC110114 Tablet; Drug: Sofosbuvir Tablet
- 1200 mg multiple doses (Experimental): Subjects receiving 1200 mg HEC110114 tablet (N=6) or sofosbuvir tablets(N=2) once daily (q.d.) for 3 days
  Interventions: Drug: Sofosbuvir Tablet

INTERVENTIONS:
Drug: HEC110114 Tablet — administered orally once daily
  Arms: 600 mg multiple doses; 800 mg multiple doses
Drug: Sofosbuvir Tablet — administered orally once daily

SUMMARY:
A Phase Ib/IIa, Single Center, Randomized, open, Sofosbuvir-controlled, Multiple Ascending Dose Study to Access the Tolerability，Pharmacokinetics and Pharmacodynamics of HEC110114 Tablets in HCV-infected Subjects

DETAILED DESCRIPTION:
A total of 24 evaluable patients will be enrolled in this study. The study randomly divided into three dose groups and HEC110114 tablets planned dose levels are 600, 800, and 1200 mg, sofosbuvir tablets planned dose levels are 400 mg .

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions;
* Be able to complete the study according to the trail protocol;
* Subjects (including partners) have no pregnancy plan within six months after the last dose of study drug and voluntarily take effective contraceptive measures;
* Male subjects and must be 18 to 65 years of age inclusive;
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive, and a body weight ≥50 kg for males and ≥45 kg for females;
* No previous treatment with any direct-acting antiviral (DAA) drugs for HCV, such as Simeprevir, Sofosbuvir, Daclatasvir etc;
* HCV RNA ≥10*5 IU/mL at screening (Roche COBAS Taqman);
* Chronic genotype 1-6 HCV Infection, multiple genotypes, subtype unidentifiable or others ;
* Serum ALT ≤5 times ULN.

Exclusion Criteria:

* Allergies constitution ( multiple drug and food allergies);
* History of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits or 100 mL of wine);
* Donation or loss of blood over 450 mL within 3 months prior to screening;
* History of any non-HCV liver diseases, including but not limited to hemochromatosis, primary biliary cirrhosis, Wilson's disease, autoimmune hepatitis, drug or alcoholic hepatitis, non-alcoholic steatohepatitis, etc;
* 12-lead ECG with clinically significant;
* Pregnant or lactating women;
* Creatinine clearance < 60 mL/min;
* Subjects deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From Days 1-10
  Incidence of adverse events

SECONDARY OUTCOMES:
Cmax | At pre-defined intervals from Days 1-7
  Maximum Observed Plasma Concentration
Tmax | At pre-defined intervals from Days 1-7
  Time to Maximum Observed Plasma Concentration
T1/2 T1/2 T1/2 T1/2 | At pre-defined intervals from Days 1-7
  Apparent Half-Life
AUClast | At pre-defined intervals from Days 1-7
  Area Under the Plasma Concentration vs Time Curve to Last Measurable Concentration
HCV RNA | At pre-defined intervals from Days 1-10
  HCV RNA declined from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Doctor, Principal Investigator — The First Hospital of Jilin University; Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Jilin, Changchun, China

IPD SHARING:
Plan to Share IPD: No